CLINICAL TRIAL: NCT06516081
Title: Efficacy of Sprinkles® and Iron Folic Acid Tablets to Control Anemia During Pregnancy
Brief Title: Controlling Anemia During Pregnancy: Sprinkles Versus IFA Tablets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Heinz Endowments (Other)
Responsible Party: Principal Investigator, Stanley Zlotkin, Chief, Global Child Health, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1000007390
Record Dates: First submitted 2021-04-14; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Anemia
Keywords: anemia; pregnancy; sprinkles; iron; folic acid
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: Iron folic acid tablets versus micronutrient powders containing iron and folic acid (Sprinkles)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Micronutrient powders (Sprinkles®). One sachet daily containing minerals and vitamins in powder form.
  Interventions: Dietary Supplement: Micronutrient powder (Sprinkles®)
- Comparator arm (Active Comparator): IFA tables daily
  Interventions: Dietary Supplement: Micronutrient powder (Sprinkles®)

INTERVENTIONS:
Dietary Supplement: Micronutrient powder (Sprinkles®)
  Other Names: Iron folic acid tablets

SUMMARY:
'Very significant progress has been made but the job is less than half done' may summarise the efforts made to control vitamin A and iodine deficiency disorders. Unfortunately, in the case of iron deficiency, the most common nutritional deficiency in the world, the story is much worse. Among the population groups mostly affected by its associated anemia are pregnant women. In clinical trials, where the intake of daily doses of iron tablets has been ensured, it was shown that this intervention can prevent anemia. However, when this intervention has been implemented in non-research settings, it has had limited effect mainly due to associated side effects and lack of motivation bringing about low compliance. New effective strategies are thus needed to deliver iron and other micronutrients that would overcome the problem of low compliance. Micronutrient powders (MNPs) (Sprinkles®) are an innovative approach that delivers necessary micronutrients including iron and folic acid during pregnancy through home-based food fortification. The objectives of the current research proposal are to provide Sprinkles or iron and folic acid tablets to pregnant women in rural Bangladesh and compare outcomes including compliance and hematological status. If Sprinkles® are determined to be equivalent or better than the traditional iron and folic acid tablets, then the next step would be to determine the effectiveness of this new intervention.

DETAILED DESCRIPTION:
Iron deficiency and anemia during pregnancy have been identified by the World Health Organization (WHO) as a priority issue. The current intervention recommended for developing countries, iron and folic acid tablets, has been shown to have low effectiveness. Alternate approaches are thus called for. It is proposed to test a new micronutrient intervention including iron and folic acid in the form of Sprinkles® to help decrease the high prevalence of iron deficiency and anemia during pregnancy. The proposed study is a cluster randomized trial to be carried out in 40 community-based antenatal care centres (ANCCs) operated by BRAC (formerly known as the Bangladesh Rural Advancement Committee), the largest non-governmental organization (NGO) in Bangladesh.

Two interventions are planned: (i) iron-folic acid (IFA) tablets; and (ii) Sprinkles®. As per guidelines set by the WHO for countries where the prevalence of anemia is > 40% (e.g. Bangladesh), 60 mg of elemental iron (as Sprinkles® or IFA tablets) will be provided to pregnant women for daily use starting at the first ANCC visit and lasting throughout the pregnancy and continued until 3 months post-partum. In addition, as per previous WHO guidelines, each tablet or Sprinkles® sachets will also contain 400μg of folic acid. For women in the IFA tablet group, one IFA tablet will be taken daily. For women in the Sprinkles® group, one sachet will be taken daily by sprinkling the entire contents of the sachet over a semi-solid food prior to consumption. Sprinkles® will contain 60 mg of elemental iron as encapsulated ferrous fumarate and 400 μg of folic acid. During the study, participants will be monitored for hematological status as well as for adherence and side effects using structured, pre-tested questionnaires.

Women will be recruited from ANCCs in the rural sub-district of Kaligonj, Bangladesh. Kaligonj has a relatively homogenous population in terms of socio-economic status, language and culture, and importantly, is located in a flood-free zone less than 50 km from Dhaka. As of December 2004, there were 100 community-based ANCCs in the Kaligonj sub-district, each operated by a trained BRAC health worker and assisted by an indigenous female community health worker (CHW). Each ANCC serves a village or a population of around 300 households. An ANCC is set up in a village for one day every month to reach all pregnant women residing in that village; thus women routinely attend the ANCC in their own village.

The inclusion criteria for the study are pregnant women, ages between 15-45 years, who have a gestational age between 14-20 weeks. For logistical reasons it is not possible to start all women at the same point. This difference in post conceptual age will be accounted for statistically. Recall of Last Menstrual Period (LMP) will approximate the gestational age in weeks; gestational age is estimated from the first day of the LMP. Therefore, any woman with gestational age > 20 weeks will be excluded. A calendar of local events will be developed to assist each of the women to recall their LMP with a greater precision. Women with Hb < 70 g/L (severely anemic according to WHO) at the start of the study will be excluded and referred to the Medical Officer at the nearest government or BRAC health centre for appropriate investigation and therapy. Women already on iron supplementation prior to the study start will not be included. Trained health workers at the ANCC will assess each potential subject for uncontrolled hypertension. Those with a known history of liver, heart or kidney disease, cancer or severe infections will be excluded. It is not possible to define all illnesses that would lead to exclusion, but generally those women requiring significant medical care, above that normally received during pregnancy will be excluded. All women must freely consent to participation.

The primary outcome is the hemoglobin (Hb) concentration. Trained nurses will collect finger-prick blood using standard techniques at 24, 28 and 32 weeks of gestation. Repeated measures are planned at specific gestational ages because a U-shaped curve of mean Hb concentrations by stage of pregnancy has been described . Hb will be measured from a drop of blood using a portable HEMOCUE B-hemoglobin photometer (HemoCue®, Angelholm, Sweden). Trained field workers will also use structured questionnaires to collect information on side effects during visits 2-7. The structured questionnaires are developed from PUQE for information on nausea and vomiting, and from previous studies which collected information on GI symptoms and stool colour, consistency and frequency. Other side effects including hospitalization, adverse events and deaths will also be collected. All forms will be pre-tested and finalized.

The sample size estimation was based on the primary outcome, the mean Hb concentrations at 24, 28 and 32nd week gestational age; the investigators assumed that the mean Hb in the iron and folic acid tablet group would be 125 g/L with a between-subject standard deviation of 15 g/L. An alpha=0.05 will be used, so that the investigators will reject H0 and declare Sprinkles® non-inferior with at most a 5% chance when it actually is inferior. Power was calculated under the hypothesis that Sprinkles® and iron and folic acid tablets are equivalent. The total sample size at follow-up is 352 and power is 91%. Loss-to-follow-up has previously been estimated at up to 35% in this population, 12 women will be recruited per ANCC to obtain, on average, around 9 women per centre with complete follow-up.

Analysis will be on an 'intention-to-treat' basis. Due to the clustered design, it may be necessary to assess comparability of baseline variables using descriptive statistics. The main outcome variable will be Hb concentrations at the 24, 28 and 32nd week of gestational age. A linear mixed-effects regression model will be used with Hb concentrations at the three post-conceptual ages as the dependent variable. The fixed effects predictors will be treatment group allocation, baseline Hb and post-conceptual age (to account for the anticipated U-shape in hemoglobin concentrations); the random effects will be subject (to account for repeated measurements) and ANCCs (to account for clustering). If the parameter for group allocation is significantly higher than -5g/L, the investigators will conclude that Sprinkles® are non-inferior to iron and folic acid tablets for the effect on hemoglobin concentrations during pregnancy.

Secondary analyses will also be conducted. The investigators will compare the PUQE scores of nausea and vomiting per woman for the two groups via random effects linear regression models (cluster as a random effect). Similar models will be used to compare episodes of GI complaints (stomach pain, heart burn) and stool pattern per woman for the two groups. Adherence, (although not an outcome) will be reported as the percentage of sachets/tablets used (after accounting for lost or shared) out of the total assigned.

Data analysts will be blinded to group assignments at all times. Since women will be recruited between 14-20 weeks of gestation, there will be some variation in length of intervention. The investigators plan to do a subgroup analysis using gestational age at the time of recruitment as a covariate and will examine its interaction with the group effect in the mixed effects linear model previously described for the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, ages between 15-45 years, who have a gestational age between 14-20 weeks

Exclusion Criteria:

* Pregnant women with Hb < 70 g/L (severely anemic according to WHO)
* Pregnant women already on iron supplementation prior to the study start
* Pregnant women with a known history of liver, heart or kidney disease, cancer or severe infections
* Pregnant women requiring significant medical care, above that normally received during pregnancy

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 480 (Actual)
Dates: Start 2005-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Hemoglobin concentration (g/L) | 24 weeks of gestation
  Hemoglobin concentration
Hemoglobin concentration (g/L) | 28 weeks of gestation
  Hemoglobin concentration
Hemoglobin concentration (g/L) | 32 weeks of gestation
  Hemoglobin concentration

SECONDARY OUTCOMES:
Adverse effects | Weekly during weeks 2-7 following study recruitment.
  Questionnaire on nausea, vomiting and GI disturbances (heartburn and 'stomach' pain) and stool pattern (consistency and colour)
Adherence . | Weekly during weeks 2-7 following study recruitment.
  Questionnaire on adherence
Acceptability of the interventions | Weekly during weeks 2-7 following study recruitment.
  Questionnaire on acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Stanley H Zlotkin, MD, PhD, Principal Investigator — The Hospital for Sick Children, Toronto, Ontario Canada
Locations (1):
- Research and Evaluation Division, BRAC, Dhaka, Bangladesh